CLINICAL TRIAL: NCT03348917
Title: The Effect of Skin Cleansers on the Skin Surface Microbiome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Manufacturing Pte Ltd. (Industry)
Collaborators: Genome Institute of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: BTD16-SG-402
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Skin Health
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Intervention Model Description: Twelve healthy volunteers will be randomized into three arms with three different treatment sequences with four healthy volunteers in each arm. Up to fifteen healthy volunteers may be recruited with the consideration that up to three subjects may drop out.
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment sequence Group 1 (Active Comparator): Treatment Sequence Group 1 = A -> B -> C
  Treatment A = Betadine® 7.5% skin cleanser (PVP-I 7.5%)
  Treatment B = 4% chlorhexidine skin cleanser - Unity antiseptic hand wash (no alcohol)
  Treatment C = Plain non antibacterial soap - Guardian gel hand wash (not medicated)
  Interventions: Drug: 7.5% Povidone-Iodine [PVP-I]; Drug: 4% chlorhexidine skin cleanser; Drug: Plain non antibacterial soap
- Treatment sequence Group 2 (Active Comparator): Treatment Sequence Group 2 = B -> C -> A
  Treatment B = 4% chlorhexidine skin cleanser - Unity antiseptic hand wash (no alcohol)
  Treatment C = Plain non antibacterial soap - Guardian gel hand wash (not medicated)
  Treatment A = Betadine® 7.5% skin cleanser (PVP-I 7.5%)
  Interventions: Drug: 7.5% Povidone-Iodine [PVP-I]; Drug: 4% chlorhexidine skin cleanser; Drug: Plain non antibacterial soap
- Treatment sequence Group 3 (Active Comparator): Treatment Sequence Group 3 = C -> A ->B
  Treatment C = Plain non antibacterial soap - Guardian gel hand wash (not medicated)
  Treatment A = Betadine® 7.5% skin cleanser (PVP-I 7.5%)
  Treatment B = 4% chlorhexidine skin cleanser - Unity antiseptic hand wash (no alcohol)
  Interventions: Drug: 7.5% Povidone-Iodine [PVP-I]; Drug: 4% chlorhexidine skin cleanser; Drug: Plain non antibacterial soap

INTERVENTIONS:
Drug: 7.5% Povidone-Iodine [PVP-I] — Betadine® 7.5% skin cleanser (PVP-I 7.5%)
Drug: 4% chlorhexidine skin cleanser — Unity antiseptic hand wash (no alcohol)
Drug: Plain non antibacterial soap — Guardian gel hand wash (not medicated),

SUMMARY:
This study determines the effects of a single application of different antiseptic skin cleansers on the composition of the skin surface microbiome using next-generation sequencing (NGS) techniques. Twelve healthy volunteers will receive all three test products in a randomized order to compare the effects of each skin cleanser.

DETAILED DESCRIPTION:
Disinfectants and oral antiseptics including PVP-I are known to kill microorganisms to a variable extent, at a variable range of time points. Microorganisms may be protected from disinfectants by production of thick masses of cells and extracellular materials, or biofilms. Moreover, antiseptics should not lead to dysbiosis after use. Dysbiosis is a negative change in the microbiome of a particular skin or mucosal region. The Human Microbiome project showed, that every area has a specific microbiota in which the human host lives with an abundance of commensal, synergistic, and potentially pathogenic microorganisms. Antiseptics with efficacy gaps and resistance may induce such dysbiosis, especially after prolonged use. It is envisaged that twelve healthy volunteers will complete the study. Each healthy volunteer will apply the test product according to a developed protocol, between established wash out periods.

The ability of the test product (Commercially available - Betadine® 7.5% skin cleanser (PVP-I 7.5%)) compared to the reference products (commercially available 4% chlorhexidine skin cleanser - Unity antiseptic hand wash (no alcohol) and Plain non antibacterial soap - Guardian gel hand wash (not medicated)) to reduce resident and transient microflora will be assessed. The hand wash products will also be assessed for their ability to maintain and/or restore balanced microflora.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between age 21 to 65 years
* Must wear short sleeved shirts/blouses during each visit
* Non-smoker
* Good general and mental health with, in the opinion of investigator or the qualified medical designee:

  1. No clinically significant and relevant abnormalities of medical history or physical examination;
  2. Absence of any condition that would impact the subject's safety or health or affect the subject's ability to understand and comply with the study procedures.
* Prepared to use the provided wash products that do not contain any antimicrobials (non antibacterial shampoo [Pantene® Pro-V], non antibacterial body wash [Dove®body wash] and non antibacterial hand wash [Guardian gel hand wash]) after providing consent and during the whole study
* Healthy and intact skin in the test area (e.g., no skin allergy, visible bleeding, skin inflammation, skin ulcer or skin lesion, no need for cutaneous treatment)
* Must have given written informed consent
* Women of child-bearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.

Exclusion Criteria:

* Women who are pregnant or have a positive urine pregnancy test or intending to become pregnant during the overall study period
* Women who are breast-feeding
* Allergy or contraindication to any test product substance (active or excipients)
* Any visible signs of skin dermatitis on the hands, e.g., eczema
* Use of anti-dandruff shampoo or any other shampoo/hand/body wash products apart from those provided, within 2 days prior to Visit 2 (Day 0) and also during the whole study
* Systemic or topical or oral antibiotic or antifungal in the past 2 months before Screening and during the study
* Medication use (e.g., lithium therapy, immunosuppressive medication, systemic or inhaled glucocorticoids) in the past 2 months before Screening and during the study
* Recent history (within the last 1 year) of alcohol or other substance abuse
* Known hyperthyroidism or other ongoing thyroid diseases
* Minor ailments such as like cough, cold, upper respiratory tract infection(s) within 2 weeks and during the study
* Any known serious ongoing disease
* Unwillingness or inability to comply with the requirements of the protocol
* Participation in any other drug, biologic, device, or clinical study or treatment with any investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) before Screening
* An employee of the sponsor or study site or their immediate family member
* Subject who has been treated with cancer within the last 1 year.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Composition of skin microbiome - reduction of microflora amount | [Time Frame: Skin Strip 1: 0 Min, Skin Strip 2: 3 min (post treatment) and Skin Strip 3: 240 min (post treatment)]
  The change in amount of skin microflora species composition from baseline after the usage of a single application of different skin cleansers using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins.
Composition of skin microbiome - maintenance of healthy microflora amount | [Time Frame: Skin Strip 1: 0 Min, Skin Strip 2: 3 min (post treatment) and Skin Strip 3: 240 min (post treatment)]
  The change in amount of healthy skin microflora species composition from baseline after the usage of a single application of different skin cleansers using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins.
Composition of skin microbiome - reduction of microflora variety | [Time Frame: Skin Strip 1: 0 Min, Skin Strip 2: 3 min (post treatment) and Skin Strip 3: 240 min (post treatment)]
  The change in variety of skin microflora species composition from baseline after the usage of a single application of different skin cleansers using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins.
Composition of skin microbiome - maintenance of healthy microflora variety | [Time Frame: Skin Strip 1: 0 Min, Skin Strip 2: 3 min (post treatment) and Skin Strip 3: 240 min (post treatment)]
  The change in variety of healthy skin microflora species composition from baseline after the usage of a single application of different skin cleansers using next generation sequencing (NGS) and real-time PCR techniques at 3 mins and 240 mins.

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Su Yien Subash Chandran, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No